CLINICAL TRIAL: NCT04233892
Title: Clinical Study of in Situ Regeneration of Endometrium
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yali Hu (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Yali Hu, Professor，Chief Physician of Obstetrics and Gynecology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC201900202
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female, of Uterine Origin; Endometrial Fibrosis
Keywords: thin endometrium; infertility
MeSH Terms: conditions — Infertility | interventions — basic fibroblast growth factor-kidney disease domain-collagen-binding domain fusion protein, mouse; Collagen; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD-bFGF (Experimental)
  Interventions: Drug: CBD-bFGF
- Collagen/BMMNCs (Experimental)
  Interventions: Drug: Collagen/BMMNCs
- Estrogen (Experimental)
  Interventions: Drug: Estrogen

INTERVENTIONS:
Drug: CBD-bFGF — CBD-bFGF will be injected into the endometrium after hysteroscopy under the guidance of ultrasound
  Arms: CBD-bFGF
Drug: Collagen/BMMNCs — A collagen scaffold loaded with BMMNCs will be transplanted into the uterine cavity after hysteroscopy under the guidance of ultrasound
  Arms: Collagen/BMMNCs
Drug: Estrogen — Patients will receive regular estrogen therapy
  Arms: Estrogen

SUMMARY:
Thin endometrium will lead to hypomenorrhea，infertility and recurrent pregnancy loss and there are few effective methods to increase the endometrial thickness and improve the fertility outcomes. Patients with thin endometrium will be divided into three groups and receive estrogen therapy, stem cell therapy and growth factor therapy respectively. This randomized controlled clinical study is carried out to explore the optimal treatment method and best indications for thin endometrium.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with thin endometrium (4mm≤ EMT <7mm )or scarred endometrium (scarred area≤70%) which is nonresponsive to estrogen stimulation 2.Infertile patients with clear fertility desires 3.20-42 years old 4.Normal ovarian function or with frozen embryos 5.Willing to participate in follow-up

Exclusion Criteria:

1. Endometrial thickness <4mm or scarred endometrial area>70%
2. Uterine cavity out of shape and the cavity depth<6.5mm
3. Abnormal chromosome karyotype
4. Uterine diseases including large intramural myomas, severe endometriosis, severe adenomyosis, severe congenital uterine malformations, endometrial tuberculosis, vaginitis and endometritis
5. Systemic diseases: hypertension, diabetes, and so on
6. Contraindications to pregnancy
7. Contraindications to hormone replacement therapy
8. Medical history of pelvic tumors or receiving pelvic radiotherapy 9 .Involved in other clinical studies

10. Unable to adhere to the follow-up

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 345 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Endometrial thickness | 6 months
  Endometrial thickness evaluated by transvaginal sonography during late proliferative phase
Ongoing pregnancy rate | 24 months
  The presence of a living intrauterine fetus on TVU at the 12th week of gestation

SECONDARY OUTCOMES:
Endometrial blood flow | 6 months
  Endometrial blood flow evaluated by transvaginal sonography
Pregnancy related complications | 24 months
  Miscarriage rate, live birth rate, ET cycle cancellation rate,Placenta related complications
Histological changes of endometrium | 12 months
  Histological changes of the thin endometrium before and after treatment
Menstrual blood volume | 6 months
  The change of menstrual blood volume after treatment compared with pre-treatment

OTHER OUTCOMES:
Adverse event rate | 24 months
  The occurrence of infections, allergies, abdominal pain, uterine perforation and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, MD,PhD, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China